CLINICAL TRIAL: NCT07159295
Title: Betreat (Xaloc1) Benralizumab Study: Retrospective, Observational Study in Portuguese Hospitals to Describe Patient Characteristics, Treatment Patterns and Outcomes
Brief Title: Study in Portuguese Hospitals to Describe Patient Characteristics, Treatment Patterns and Outcomes
Acronym: Betreat
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00088
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Benralizumab is indicated as an add-on maintenance treatment in adult patients with severe eosinophilic asthma inadequately controlled despite high-dose inhaled corticosteroids plus long-acting β2-agonists. It has been reimbursed in Portugal as an add-on therapy since May 2019. In order of this, there is crucial need in Portugal to provide key real-word evidence on benralizumab therapy.

DETAILED DESCRIPTION:
This is a real-world retrospective, multicentric, observational study, utilizing secondary data collection from medical records of adults patients (≥18 years) with severe asthma (maintenance treatment with high dose inhaled corticosteroids combined with long-acting agonist β2) and eosinophilic phenotype, who, at the discretion of the physician, received benralizumab accordingly to the clinical practice, in the period after the marketing authorization of benralizumab.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with severe asthma treated with benralizumab, who had their first benralizumab dose between July 2019 and October 2020

  * Patients who have at least 1 benralizumab injection and with at least 3 months follow-up data from the first injection.
  * Give voluntary signed informed consent

Exclusion Criteria:

* Currently receiving benralizumab or any other biologic drug for the treatment of asthma in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe eosinophilic asthma patients aged 18 and above, treated with benralizumab and who have had their first benralizumab dose between July 2019 and October 2020 and who have at least 1 benralizumab injection and with at least 3 months follow-up data from the first injection.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Baseline demographic and clinical characteristics of severe eosinophilic asthma patients treated with benralizumab | Baseline/Index date
  Demographic: Gender, age, BMI, smoking history Clinical: age of asthma diagnosis, ACT score, CARAT score, blood eosinophil count, FeNO, Lung function, FVC, Reversibility of FEV1, Total IgE in peripheral blood, Skin PRICK test
Background treatment patterns of severe eosinophilic asthma patients at baseline and after benralizumab initiation and treatment duration with benralizumab | Baseline, 3, 6, 12 and 24 months
  Medication history: asthma treatment type, doses and treatment duration Proportion of patients with biologic discontinued and reason for discontinuation Benralizumab treatment patterns: benralizumab treatment duration, frequency of benralizumab treatment discontinuation, time to treatment discontinuation and frequency and type of concurrent respiratory medication

SECONDARY OUTCOMES:
Clinical outcomes after initiation of benralizumab theraoy in severe eosinophilic asthma patients | Baseline, 3, 6, 12 and 24 months
  Frequency of asthma exacerbations, annual rate of severe exacerbation, mean change in lung function (FEV1), FVC, reversibility of FEV1, blood eosinophil count, FeNO, Total IgE in peripheral blood, CARAT and ACT scores, proportion of patients achieving an improvement in CARAT ACT, percentage of patients with OCS ≤5mg/day, percentage change in daily OCS dose, percentage of patients experiencing reduction daily OCS use from index date by >0%, ≥25%, ≥50%, ≥75%, ≥90% and 100%
Asthma-related Healthcare resource utilization (HCRU) among severe eosinophilic asthma patients before and after initiation of benralizumab therapy | Baseline, 3, 6, 12 and 24 months
  Number of emergency room visits, Number of schedule medical visits for asthma, Number of unscheduled medical visits for asthma, Number of hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Fernandes, Principal Investigator — Hospital Pedro Hispano; Claudia Loureiro, Principal Investigator — CHUC Pneumo; Carlos Loureiro, Principal Investigator — CHUC Imuno; Ulisses Brito, Principal Investigator — CHUA - Faro; Inês Belchior, Principal Investigator — CHUA - Portimão; Ana Mendes, Principal Investigator — CHLN- HSM - Imuno; Gonçalo Portugal, Principal Investigator — CHLN - HSM - Pneumo; Rita Boaventura, Principal Investigator — Hospital S. João- Pneumo; José Plácido, Principal Investigator — Hospital S. João - Imuno; Cecília Pardal, Principal Investigator — Hospital Prof. Dr. Fernando Fonseca; Gustavo Reis, Principal Investigator — Hospital Distrital de Santarém; Ricardo Lima, Principal Investigator — CHVNGE; Liliana Ribeiro, Principal Investigator — Hospital Centre Hospitalar de Trás-os-Montes e Alto Douro; Nuno Pires, Principal Investigator — HSMM- Barcelos; Nuno Sousa, Principal Investigator — Hospital Leiria; Filipa Carriço, Principal Investigator — Hospital São João - CRI
Locations (16):
- Portugal (16):
  - Hospital Prof. Dr. Fernando Fonseca, Amadora
  - HSMM, Barcelos
  - CHUC - Imunoalergologia, Coimbra
  - CHUC - Pneumologia, Coimbra
  - CHUA, Faro
  - Hospital Leiria, Leiria
  - Chln - Hsm, Lisbon
  - Chuln - Hsm, Lisbon
  - Hospital Pedro Hispano, Matosinhos Municipality
  - CHUA, Portimão
  - CHUSJ - Imuno, Porto
  - CHUSJ - Pneumo, Porto
  - Chusj - Cri, Porto
  - Hospital Distrital de Santarém, Santarém
  - CHVNGE, Vila Nova de Gaia
  - CHTMAD, Vila Real

IPD SHARING:
Plan to Share IPD: No
No IPD is planned to be shared.

REFERENCES:
- See also: D3250R00088_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00088&attachmentIdentifier=1aa77882-f9af-4dfc-92f4-f8cc413a6053&fileName=D3250R00088_CSR_Synopsis_Redacted.pdf&versionIdentifier=